CLINICAL TRIAL: NCT06065709
Title: The Effect of Mindfulness Breath Awareness Meditation on Health Profile, Vital Signs, and Fetal Heart Rate in Pregnant Women Diagnosed With Preeclampsia
Brief Title: Mindfulness Breath Awareness Meditation and Preeclampsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Kilicli (Other)
Responsible Party: Sponsor-Investigator, Aysegul Kilicli, gaziantep university health sciences enstitute nursing department PhD, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MEDITATION AND PREECLAMPSİA
Record Dates: First submitted 2023-09-19; First posted 2023-10-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Mindfulness Breath Awareness Meditation; Preeclampsia
Keywords: Mindfulness breath awareness meditation; Preeclampsia; Pregnant women; Health profile; Vital signs; Fetal heart rate
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness breath awareness meditation group (Experimental): Mindfulness breath awareness meditation will be performed nine times in total, once every eight hours within 72 hours, to the pregnant woman who is hospitalised in the perinatology service of the hospital with the diagnosis of preeclampsia. Each session will last 30 minutes.
  A 4-stage mindfulness breath awareness meditation includes the following stages:
  Stage 1 - Body Harmony. Stage 2 - Counting as you Exhale Stage 3 - Counting while Breathing Stage 4 - Sit Still and Witness.
  Interventions: Behavioral: Mindfulness breath awareness meditation
- control group (No Intervention): only mindfulness breath awareness meditation will not be applied to the control group.

INTERVENTIONS:
Behavioral: Mindfulness breath awareness meditation — Mindfulness breath awareness meditation
  Arms: Mindfulness breath awareness meditation group

SUMMARY:
The effect of mindfulness breath awareness meditation on health profile, vital signs, and fetal heart rate in pregnant women with preeclampsia

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of mindfulness breath awareness meditation (MBAM) on health profile, vital signs, and fetal heart rate in pregnant women with preeclampsia.

Sample size:

* There will be two groups in the study.
* Experiment group is breath awareness meditation group.
* The sample size of the study is 66 women.
* The sample size will be divided into two and 33 women will be randomly assigned to each group.

Application time:

* The application will be started after the pregnant women diagnosed with pre-eclampsia is admitted to the Perinatology service.
* It will be applied total nine times in once every eight hours during the 72 hours that the pregnant women diagnosed with 20 minutes.
* Only mindfulness breath awareness meditation (MBAM) will not be applied to the control group. Care and follow-up will be performed in parallel with the individuals in the experimental group.

Data Collection Tools:

* Descriptive Information Form
* Nottingham Health Profile Scale

Measurement time:

* Pregnant women will fill in the Introductory Information Form before the first application.
* Each session of mindfulness breath awareness meditation practice will 20 minutes.
* Pregnant women will fill the Nottingham Health Profile Scale before the first application. It will then be refilled at the same time every 24 hours for 72 hours. The Nottingham Health Profile will be completed a total of four times.
* Vital signs (systolic and diastolic blood pressure, body temperature, pulse, respiration, oxygen saturation) will be measured immediately before the first application. They will then be refilled at the same time every 24 hours for 72 hours. Vital signs will be completed a total of four times.
* Fetal heart rate and fetal movement count will be measured immediately before the first application. They will then be refilled at the same time every 24 hours for 72 hours. Fetal heart rate and fetal movement count will be assessed by Non-stress Testing (NST). The pregnant woman will undergo NST for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who is admitted to the Perinatology Service of the hospital with the diagnosis of preeclampsia,
* who is 19 to 49 years old,
* who is 20 and over weeks of gestation,
* who followes by at least three days of hospitalization in the ward.

Exclusion Criteria:

* Pregnant women who do not meet the inclusion criteria and who voluntarily withdraw at any stage after inclusion will be excluded from the study.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women diagnosed with preeclampsia
Enrollment: 66 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Nottingham Health Profile | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Nottingham Health Profile The scale consists of 38 questions and 6 sub-dimensions. The scale consists of 8 questions on physical activity (PA), 8 questions on pain (P), 5 questions on sleep (S), 3 questions on energy level (EL), 9 questions on emotional reactions (ER), 5 questions on social isolation (SI). Questions are answered as 'yes' or 'no', item score calculations in each sub-dimension differ, the best score that can be obtained from each sub-dimension is '0' and the worst score is '100'. The minimum score that can be obtained from the whole scale is 0 and the maximum score is 600. Quality of life improves as the score decreases.
Fetal heart rate | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Fetal heart rate
Body temperature | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Body temperature
Pulse | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Pulse
Systolic blood pressure | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Systolic blood pressure
Diastolic blood pressure | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Diastolic blood pressure
Respiratory rate | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Respiratory rate
Oxygen saturation | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Oxygen saturation

SECONDARY OUTCOMES:
fetal movement count | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  fetal movement count
Nottingham Health Profile subdimensions | It will be evaluated before the first application and then every 24 hours for a total of 4 times
  Nottingham Health Profile subdimensions physical activity, pain, sleep, energy, emotional reactions, and social isolation

CONTACTS AND LOCATIONS:
Locations (1):
- Şanlıurfa training and research hospital, Sanliurfa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No